CLINICAL TRIAL: NCT00275834
Title: Zonisamide for Weight Reduction in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00005514; R01DK067352 (NIH); 1R01DK067352 (NIH)
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: obesity treatment; weight loss; antiobesity drugs; zonisamide
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Zonisamide 400 mg
  Interventions: Drug: Zonisamide
- B (Experimental): Zonisamide 200 mg
  Interventions: Drug: Zonisamide
- C (Placebo Comparator): matching placebo
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — zonisamide 400 mg, 200 mg, or placebo

SUMMARY:
The primary aim of this study is to assess long-term weight loss efficacy of zonisamide relative to placebo in obese patients prescribed a dietary intervention.

DETAILED DESCRIPTION:
This RCT compares two doses of zonisamide and placebo for one year. A total of 225 subjects are randomly assigned to one of the three treatment interventions at Duke University Medical Centre. The primary outcome measure is change in body weight in kilograms. Secondary outcomes include changes in waist circumference, glycaemic and inflammatory markers, lipids, food craving, hunger and satiety, quality of life, blood pressure and heart rate.

ELIGIBILITY:
Inclusion Criteria: Age 18-65 years; BMI 30-50

Exclusion Criteria:

Secondary obesity; Significant cardiovascular disease; Stroke, seizure disorder or other significant neurological disease; Significant liver or gallbladder disease; Significant renal disease or history of kidney stones; HIV positive status; Diabetes mellitus; Untreated or unstable hypothyroidism Malignancy in the past 5 years; Concomitant medications that cause significant weight gain or weight loss; Concomitant use of prescription or OTC weight loss medications; Had bariatric surgery or planning surgery in the next 1 year; Weight change of more than 4 kg in the past 3 months; Suicidal subjects; Major depression in the past 6 months; History of psychosis, bipolar disorder, or severe personality disorders; Subjects taking antipsychotics or mood stabilisers; Alcohol or substance abuse in the past 6 months; Currently taking zonisamide or other antiepileptic drugs; History of hypersensitivity to zonisamide or sulfonamides; Pregnant or planning pregnancy in the next year, or breastfeeding; Severe physical disability; Current participation in a commercial weight loss program or planning to participate; Currently following low-carbohydrate, high protein, high fat diet; Use of investigational medications or devices (current or past 4 weeks)

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2006-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kishore M Gadde, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Centre, Durham, North Carolina, United States

REFERENCES:
- [Background] Gadde KM, Kopping MF, Wagner HR 2nd, Yonish GM, Allison DB, Bray GA. Zonisamide for weight reduction in obese adults: a 1-year randomized controlled trial. Arch Intern Med. 2012 Nov 12;172(20):1557-64. doi: 10.1001/2013.jamainternmed.99. PMID 23147455
- [Derived] Shin JH, Gadde KM, Ostbye T, Bray GA. Weight changes in obese adults 6-months after discontinuation of double-blind zonisamide or placebo treatment. Diabetes Obes Metab. 2014 Aug;16(8):766-8. doi: 10.1111/dom.12275. Epub 2014 Mar 10. PMID 25123600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Duke University Medical Center between 2006 and 2011.
Pre-assignment Details: Participants are considered to have completed the study if they returned for final study visit. The number completed represents participants who stayed on study drug during the trial plus participants who discontinued study drug during the trial but continued to be followed by study team and completed the final visit assessments.
Groups:
- Placebo: Zonisamide 100 mg and placebo capsules were prepared in accordance with Good Manufacturing Practice (GMP) guidelines in Duke Compounding Facility with active pharmaceutical ingredient (Sochinaz SA, Switzerland, distributed by Bachem Americas, King of Prussia, Pennsylvania) plus dextrose as an inactive ingredient. Identical-looking placebo capsules contained dextrose.
  Each capsule contained zonisamide 100 mg or placebo, with patients and study staff blinded to contents. Dose was gradually titrated upward as follows: 1 capsule for 15 days, 2 during days 16-30, 3 capsules during days 31-45, and 4 from day 46 onward. The entire dose was taken at night. Blinded dose reduction was allowed and dose increase could be withheld. Patients had the option to discontinue the drug and remain in the study receiving only diet and lifestyle counseling.
- Zonisamide 200 mg: Dosing of matching placebo was identical.
Period: Overall Study
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Started | 74 | 76 | 75
Completed Study While on Study Drug | 54 | 51 | 62
Completed | 71 | 73 | 74
Not Completed | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg | Total
Number analyzed (Participants) | 74 | 76 | 75 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 74 | 76 | 75 | 225
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.3) | 44.2 (10.1) | 42.3 (10.0) | 43.4 (10.1)
Gender [Count of Participants; unit: Participants]
  Female | 44 | 45 | 45 | 134
  Male | 30 | 31 | 30 | 91
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 75 | 225

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: The primary endpoint was weight loss at 1-year, Month-12 weight minus baseline weight, in kilograms.
Time Frame: 1 year
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
kg | -4.0 [-5.8 to -2.3] | -4.4 [-6.1 to -2.6] | -7.3 [-9.0 to -5.6]

2. Secondary Outcome: Proportions of Patients With 5% Weight Loss
Description: These were the proportions of patients losing 5% or more weight at 1-year relative to baseline. The measures were modeled with logistic regressions that included the three-level group proxy and a baseline weight covariate.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
participants | 23 | 26 | 41

3. Secondary Outcome: Proportions of Patients With 10% Weight Loss
Description: This outcomes measure followed the same principles at measurement of proportions of patients with 5% weight loss described elsewhere.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
participants | 6 | 17 | 24

4. Secondary Outcome: Waist Circumference
Description: Analyses was based on intent-to-treat ANCOVA. Difference scores from baseline to endpoint (Month-12) for each measure were regressed on the three-level proxy denoting group while controlling for the baseline value of the same measure. Contrasts were subsequently estimated in models, which had a significant overall treatment effect.
Time Frame: 1 year
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
cm | -4.8 [-6.6 to -3.1] | -6.1 [-7.8 to -4.3] | -8.5 [-10.2 to -6.8]

5. Secondary Outcome: Inflammatory Markers (CRP)
Description: C reactive Protein (CRP)
Time Frame: 1 year
Population: Participants who had CRP testing completed
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 73 | 75 | 75
mg/L | 0.523 (0.064) | 0.536 (0.06) | 0.443 (0.044)

6. Secondary Outcome: Change in Lipids
Time Frame: baseline, 1 year
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
mg/dL
  Total Cholesterol | -1.9 [-7.2 to 3.4] | 4.1 [-1.0 to 9.2] | -0.1 [-5.0 to 4.9]
  LDL Cholesterol | -2.0 [-6.7 to 2.7] | 1.7 [-2.8 to 6.3] | -0.3 [-4.7 to 4.1]
  HDL Cholesterol | 2.5 [0.7 to 4.3] | 1.5 [-0.3 to 3.2] | 3.4 [1.7 to 5.1]
  Triglycerides | -11.3 [-22.6 to 0.0] | 0.7 [-10.1 to 11.5] | -11.7 [-22.2 to -1.1]

7. Secondary Outcome: Quality of Life as Measured by HADS_D
Description: Hospital Anxiety and Depression Scale - Depression (HADS-D) The HADS is a 14-item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale consists of 7 statements and the participant responds as to how each item applies to him/her over the past week on 4-point response scale. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: 1 year
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
units on a scale | 2.12 [1.54 to 2.70] | 2.76 [2.18 to 3.33] | 1.95 [1.38 to 2.53]

8. Secondary Outcome: Change in Blood Pressure
Time Frame: Baseline, 1 year
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Number analyzed (Participants) | 74 | 76 | 75
mm Hg
  Systolic | -0.6 [-2.9 to 1.6] | -4.4 [-6.7 to -2.1] | -1.9 [-4.1 to 0.4]
  Diastolic | -1.5 [-3.2 to 0.1] | -3.6 [-5.3 to -2.0] | -3.9 [-5.5 to -2.3]

ADVERSE EVENTS:
Time Frame: 1-year
Arm/Group | Placebo | Zonisamide 200 mg | Zonisamide 400 mg
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 30/74 | 37/76 | 39/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Zonisamide 200 mg (N=76) | Zonisamide 400 mg (N=75)
Altered taste (Gastrointestinal disorders) | 0 | 4 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 1
Nausea/vomiting (Gastrointestinal disorders) | 4 | 4 | 10
Anxiety related (Psychiatric disorders) | 2 | 5 | 7
Depression related (Psychiatric disorders) | 3 | 3 | 5
Impaired concentration (Nervous system disorders) | 1 | 1 | 4
Impaired memory (Nervous system disorders) | 1 | 5 | 8
Headache (Nervous system disorders) | 5 | 8 | 14
Fatigue (Nervous system disorders) | 2 | 4 | 7
Somnolence (Nervous system disorders) | 3 | 9 | 6
Musculoskeletal problems (Musculoskeletal and connective tissue disorders) | 9 | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No